CLINICAL TRIAL: NCT07245485
Title: Fluid Responsiveness in Coronary Artery Bypass Surgery: The Role of Carotid Artery Ultrasound and Passive Leg Raising Maneuver
Brief Title: Fluid Responsiveness With Passive Leg Raising in Patients Undergoing Coronary Artery Bypass Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: TABED 1-25-1556
Record Dates: First submitted 2025-09-24; First posted 2025-11-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Fluid Responsiveness; Passive Leg Raising; Corrected Carotid Flow Time
Keywords: Hemodynamic Monitoring; Corrected Carotid Flow Time; Passive Leg Raising

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: After the patient is placed in a 45-degree head-up position, ccFT will be measured and hemodynamic parameters will be recorded.After passive leg raising, ccFT and hemodynamic parameters will be recorded.

SUMMARY:
The aim of this study is to investigate the reliability of corrected carotid flow time (ccFT) and the percentage change in peak flow velocity (ΔVpeak), as non-invasive methods for assessing fluid responsiveness using the passive leg raising (PLR) test in patients undergoing coronary bypass surgery.

DETAILED DESCRIPTION:
This study is a single-center, prospective, and observational research. After obtaining approval from the ethics committee, 50 patients scheduled for elective coronary artery bypass surgery under general anesthesia at the Cardiovascular Surgery operating room of the Ministry of Health Ankara City Hospital will be included in the study. The study is designed as a single-center, prospective, and observational trial.

Patient data including weight, height, age, gender, BMI (body mass index), ASA classification, left ventricular ejection fraction, comorbidities, and medications will be recorded. Anesthesia induction and management will be performed in accordance with the routine practice of the anesthesia clinic. After the patient is brought to the operating table, in addition to standard hemodynamic monitoring with non-invasive blood pressure (NIBP), 5-lead ECG, and pulse oximetry, bispectral index (BIS), body temperature, and cardiac output monitoring with the Pulsion Flex device will be performed. Parameters measured by the Pulsion Flex device (CI, SVI, SVRI, SVV, PPV, DO2I, dPmx) will be recorded before and after anesthesia induction. General anesthesia will be induced with preoxygenation followed by 0.05 mg/kg midazolam, 1 mg/kg lidocaine, 3 mcg/kg fentanyl, and 2 mg/kg propofol. Muscle relaxation will be achieved with 0.6-0.8 mg/kg rocuronium, and orotracheal intubation will be performed with an appropriate tube. The target BIS value will be maintained within 40-60, and anesthesia will be maintained by adjusting the concentration of volatile anesthetics and remifentanil infusion dose (0.05-0.2 mcg/kg/min) according to hemodynamic parameters.

Ventilation mode and parameters will be set as follows: tidal volume 8 ml/kg based on ideal body weight, respiratory rate adjusted to maintain end-tidal CO₂ between 30-40 mmHg, inspiration/expiration ratio 1:2, positive end-expiratory pressure (PEEP) 5 cmH₂O, and FiO₂ 50%. After Allen's test is performed, radial artery catheterization of the non-dominant hand will be performed for invasive blood pressure monitoring, and a 7 Fr triple-lumen central venous catheter will be inserted into the right internal jugular vein for central venous pressure (CVP) monitoring. These procedures are routinely performed in patients scheduled for open thoracic surgery in our clinic. Preferably, two large-bore peripheral intravenous lines will also be inserted. Measurements will begin once patient preparation is complete, during a hemodynamically stable period, and when spontaneous respiratory effort is absent.

After the patient is placed in a 45-degree head-up semi-sitting position, hemodynamic parameters will be recorded: heart rate (HR, beats/min), systolic arterial pressure (SAP, mmHg), diastolic arterial pressure (DAP, mmHg), mean arterial pressure (MAP, mmHg), stroke volume index (SVI), cardiac index (CI), PPV, and SVV. Corrected carotid flow time (ccFT) and the percentage change in peak velocity (ΔVpeak), measured using Doppler ultrasound, will also be recorded. Ultrasound measurements will be performed with a 4-12 MHz linear probe in vascular mode. With the patient's head tilted 30 degrees to the left, a longitudinal view of the right common carotid artery will be obtained below the lower border of the thyroid cartilage, and measurements will be taken 2 cm proximal to the carotid bifurcation. Doppler will be activated, and the sample volume will be placed at an angle less than 60 degrees in the region with optimal color flow. Flow time will be measured from the beginning of the systolic upstroke to the dicrotic notch.

After one minute of passive leg raising (PLR), hemodynamic parameters as well as ccFT and ΔVpeak will be measured again and recorded. Patients demonstrating a ≥10% increase in CI measured by the Pulsion Flex device after PLR will be classified as fluid responsive, while those without such an increase will be classified as non-responders. The differences in ccFT and ΔVpeak parameters between the two groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

A total of 50 patients undergoing elective coronary artery bypass surgery under general anesthesia in the Cardiovascular Surgery operating room of the Ministry of Health Ankara Bilkent City Hospital will be included in the study.

The volunteers to be included will be patients aged between 18 and 80 years, evaluated as ASA class II-III according to the American Society of Anesthesiologists (ASA) classification.

Exclusion Criteria:

Patients who do not wish to participate in the study

Patients younger than 18 or older than 80 years

Patients with an ASA score greater than III

Patients with BMI > 35

Patients with EF < 40%

Patients with atrial fibrillation

Patients with severe valvular stenosis or insufficiency

Patients with right ventricular dysfunction

Patients with carotid artery stenosis

Patients with a history of cerebrovascular accident or transient ischemic attack

Patients with increased intra-abdominal or intracranial pressure

Patients with glaucoma

Patients with severe renal or hepatic disease

Patients who develop hemodynamic instability during the perioperative period

Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 patients undergoing elective coronary artery bypass surgery under general anesthesia in the Cardiovascular Surgery operating room
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
hemodynamic parameters (T0) | before anesthesia induction
  After patient monitoring, hemodynamic parameter values will be recorded before anesthesia induction
hemodynamic parameters (T1) | after anesthesia induction
  Hemodynamic parameters will be recorded after anesthesia induction.
ccFT and Hemodynamic parameters (T3) | After the patient is placed in a 45-degree head-up position
  After the patient is placed in a 45-degree head-up position, ccFT will be measured and hemodynamic parameters will be recorded.
ccFT and Hemodynamic Parameters (T4) | After passive leg raising
  After passive leg raising, ccFT and hemodynamic parameters will be recorded.

SECONDARY OUTCOMES:
Delta Vpeak | After the patient is placed in a 45-degree head-up position
  calculation of Delta Vpeak
Delta Vpeak | After passive leg raising
  calculation of Delta Vpeak

CONTACTS AND LOCATIONS:
Overall Officials: Ümit Karadeniz, Professor, Study Director — Ankara Bilkent City Hospital Department of Anesthesiology and Reanimation, Ankara, Çankaya
Locations (1):
- Ankara Bilkent City Hospital Department of Anesthesiology and Reanimation, Ankara, Çankaya, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singla D, Gupta B, Varshney P, Mangla M, Walikar BN, Jamir T. Role of carotid corrected flow time and peak velocity variation in predicting fluid responsiveness: a systematic review and meta-analysis. Korean J Anesthesiol. 2023 Jun;76(3):183-193. doi: 10.4097/kja.22385. Epub 2022 Nov 15. PMID 36377330
- [Background] Walker SCD, Lipszyc AC, Kilmurray M, Wilding H, Akhlaghi H. Questioning the Role of Carotid Artery Ultrasound in Assessing Fluid Responsiveness in Critical Illness: A Systematic Review and Meta-Analysis. Crit Care Res Pract. 2024 Apr 27;2024:9102961. doi: 10.1155/2024/9102961. eCollection 2024. PMID 38716052
- [Background] Cheong I, Otero Castro V, Sosa FA, Tort Oribe B, Fruchtenicht MF, Tamagnone FM, Merlo PM. Passive leg raising test using the carotid flow velocity-time integral to predict fluid responsiveness. J Ultrasound. 2024 Mar;27(1):97-104. doi: 10.1007/s40477-023-00824-1. Epub 2023 Sep 5. PMID 37668901
- [Background] Suresh V, Sethuraman M, Karunakaran J, Koshy T. Fluid responsiveness to passive leg raising in patients with and without coronary artery disease: A prospective observational study. Ann Card Anaesth. 2020 Oct-Dec;23(4):439-446. doi: 10.4103/aca.ACA_73_19. PMID 33109801